CLINICAL TRIAL: NCT04644614
Title: Effectiveness of Magnetic Stimulation in Patients With Urinary Incontinence After Radical Prostatectomy: a Prospective Randomized Sham Controlled Clinical Study
Brief Title: Pelvic Floor Magnetic Stimulation in Men With Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, PAU, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 60116787-020/38072
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Urinary Incontinence Episodes After the Magnetic Stimulation in Men With Radical Prostatectomy
Keywords: urinary incontinence; radical prostatectomy; magnetic stimulation
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Magnetic Stimulation (Active Comparator): Patients will be instructed to sit in a magnetic coil chair. Magnetic flux is generated in this field. This current stimulates the nerve or muscle of the pelvic floor. To administer MS, a stimulation amplitude of 200 μs and a repetition of 10 Hz for 10 minutes, 2 minutes rest in between, 50 Hz for 10 minutes (20 minutes total), 5 seconds on / 5 seconds off, in accordance with device literature will be adjusted to produce maximum stimuli with the cycle. During each treatment session, the device will be adjusted to receive patients the current intensity gradually increasing, reaching the maximum stimulation intensity.
  Interventions: Device: Magnetic Stimulation - Armchair type
- Group 2: Sham Magnetic Stimulation (Sham Comparator): The Sham MS treatment program will be the same as active MS in terms of duration, frequency, current duration, current intensity and general patient experience. The same magnetic chair will be used for both groups. Sham therapy application will be applied by the coordinator of the study by placing a thin deflector lead / aluminum coated plate on the magnetic coil of the magnetic chair that prevents the magnetic flux from penetrating into the patient.
  During both applications, the patients will be exposed to the same sound, vibration sensation and lighting of the device.
  Interventions: Device: Magnetic Stimulation - Armchair type

INTERVENTIONS:
Device: Magnetic Stimulation - Armchair type — MS and Sham MS will be applied two days a week, 20 minutes a day, for 8 weeks, a total of 16 sessions.
  Other Names: NovaMag NT-60

SUMMARY:
MS is a technology developed to non-invasively stimulate the central and peripheral nervous system, is applied in the treatment of UI. The MS technique aims to directly stimulate the pelvic floor muscles and sacral roots in the treatment of UI (3,4).

MS is a more acceptable, relatively painless, non-invasive and suitable electrical treatment method for patients with UI (5).

Data from studies suggest that MS may be beneficial for patients with UI after RP (1,2,5,6,7). In the literature, there are only 3 randomized controlled trials evaluating MS efficacy using a magnetic chair in patients with UI after RP (1,6,8) and one of them was published in Korean (6) and two of them in English(1,8). In these studies, MS was compared with pelvic floor muscle exercises (PFME) or electrical stimulation (ES) (intra-anal).Yokoyama et al.reported that MS and ES treatments had shown to provide earlier continence compared to the control group after RP. MS and ES are recommended as options for patients who want rapid recovery of postoperative UI(1).

Liu et al reported that MS was more effective than PTKE on incontinence symptoms and quality of life (8). However, as far as we know, there is no prospective randomized sham-controlled study evaluating the effectiveness of MS in patients with post-RP UI. In addition, there are no suggestions regarding MS in the guidelines on urinary incontinence management due to insufficient data (9). In this study, sham-controlled efficacy of MS will be evaluated in patients with UI after RP.

Our study is the first prospective randomized controlled trial comparing MS and Sham MS efficacy in patients with UI after RP. In this study, we aimed to evaluate the effectiveness of MS on incontinence related clinical parameters, quality of life, sexual functions, depression and anxiety in patients with UI after RP.

DETAILED DESCRIPTION:
This study is a prospective randomized sham-controlled study. The research will be carried out between January 2021 and June 2022 in XXX Physical Medicine and Rehabilitation (PMR) Department Urogynecological Rehabilitation Unit.

After the approval of XXX Faculty of Medicine Ethics Committee, 40 patients who admitted to XXX PMR Polyclinic with RP complaints after UI and who accepted the inclusion criteria directed to the Urogynecological Rehabilitation Unit, will be included in the study.

Patients will be informed about the content, purpose and application of the study and their written consent will be obtained.

Treatment Protocol 40 men with UI after RP who meet the exclusion and inclusion criteria will be divided into 2 groups using a table of random numbers. MS will be applied to the first group and sham MS will be applied to the second group.

Group 1: Magnetic stimulation (Active MS) Group 2: Sham MS

Group 1: Magnetic stimulation (Active MS)

Patients will be instructed to sit in a magnetic coil chair. Magnetic flux is generated in this field. This current stimulates the nerve or muscle of the pelvic floor. To administer MS, a stimulation amplitude of 200 μs and a repetition of 10 Hz for 10 minutes, 2 minutes rest in between, 50 Hz for 10 minutes (20 minutes total), 5 seconds on / 5 seconds off, in accordance with device literature will be adjusted to produce maximum stimuli with the cycle. During each treatment session, the device will be adjusted to receive patients the current intensity gradually increasing, reaching the maximum stimulation intensity. MS will be applied two days a week, 20 minutes a day, for 8 weeks, a total of 16 sessions.

Group 2: Sham MS

The Sham MS treatment program will be the same as active MS in terms of duration, frequency, current duration, current intensity and general patient experience. The same magnetic chair will be used for both groups. Sham therapy application will be applied by the coordinator of the study by placing a thin deflector lead / aluminum coated plate on the magnetic coil of the magnetic chair that prevents the magnetic flux from penetrating into the patient.

During both applications, the patients will be exposed to the same sound, vibration sensation and lighting of the device.

Patients who did not attend even one of the 16 sessions (MS and sham MS sessions) during the study period will be excluded from the study. Until the study is completed, patients will not be informed of what treatment they received. At the end of the treatment, patients in the sham group will be allowed to receive active MS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Men with RP with incontinence over ≥50 g / 24 hours
3. Patients within 1 month to 1 year after catheter removal
4. Willingness to complete and do the quality of life scale
5. Understanding procedures, benefits, and possible side effects
6. Being able to give written, informed consent

Exclusion Criteria:

1. History of conservative treatment after RP including MS
2. Previous urological surgery history
3. UI history before RP
4. Transurethral resection of the prostate due to benign prostatic hyperplasia
5. Patients receiving radiotherapy
6. Presence of urinary tract infection
7. Heart failure, presence of a pacemaker, implanted defibrillator
8. Continuing treatment for arrhythmias
9. Undiagnosed lower abdominal pain
10. Electronic device or metallic implant applied to the areas between the lumbar region and lower extremities
11. Use of drugs that may affect bladder function (antimuscarinic, duloxetine, tricyclic antidepressant, etc.)
12. History of neurogenic bladder, peripheral or central neurological pathology

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with urinary incontinence after radical prostatectomy
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Incontinence episodes | 6 weeks
  Patients with a 50% or greater reduction in incontinence episodes were consider improvement

SECONDARY OUTCOMES:
Severity of incontinence | 6 weeks
  The 24-hour pad test was carried out to evaluate urinary loss.
Three-day Bladder Diary | 6 weeks
  It was used "frequency of voiding", "incontinence episodes", "nocturia", "number of pads" from data collected with a 3-day bladder diary.
Quality of Life - Incontinence Impact Questionnaire (IIQ-7) | 6 weeks
  The IIQ-7 scale which has great validity in studies was used to assess the patient's QoL associated with incontinence problem
Level of sexual function - International Index of Erectile Function (IIEF) | 6 weeks
  Sexual functions
Level of Anxiety and Depression - Hospital Anxiety and Depression Scale (HAD) | 6 weeks
  Anxiety and Depression
Treatment satisfaction - Likert scale (1-5 ) | 6 weeks
  The patients evaluated the change of their urinary incontinence on a 5-point Likert scale (5, very satisfied; 4, satisfied; 3, equally satisfied and unsatisfied; 2, unsatisfied; 1, very unsatisfied)
Treatment Success (Continence rate) | 6 weeks
  Patients with ≤8 gr in 24-hour pad test measurement will be considered "continent"
Cure (Dry) and Improvement Rate | 6 weeks
  the absence of will be evaluated as "dryness".

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Yildiz, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unal B, Sarsan A, Yildiz N, Alkan H. Efficacy of Magnetic Stimulation in Men With Urinary Incontinence After Radical Prostatectomy: A Randomized, Quadruple-Blind, Sham-Controlled Clinical Trial. Neurourol Urodyn. 2025 Jun;44(5):1140-1148. doi: 10.1002/nau.70055. Epub 2025 Apr 14. PMID 40223765
- Available data/document: Study Protocol — https://doi.org/10.1016/j.urols.2015.06.286